CLINICAL TRIAL: NCT06266208
Title: Utility of High-resolution Ultrasound to Evaluate Dorsal Osteophyte Associated With Onychocryptosis: Correlation With Radiology.
Brief Title: Utility of High-resolution Ultrasound to Evaluate Dorsal Osteophyte
Status: Completed | Type: Observational
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Other Study IDs: UCV/2021-2022/201
Record Dates: First submitted 2024-01-25; First posted 2024-02-20 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Exostosis
Keywords: Dorsal osteophyte; Ultrasound; Nail curvature; Nail-phalanx distance
MeSH Terms: conditions — Exostoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (non-operated):: This group will consist of patients with clinical and radiological diagnosis of painful claw nail with wide nail curvature and presence of dorsal osteophyte on radiograph. They will not have received previous surgery for this condition. They will be followed up conservatively for 1 month, with baseline measurements of nail curvature, nail thickness, osteophyte height and nail-phalange distance. This group will allow correlating the osteophyte height with the degree of nail deformity without surgical intervention.
  Interventions: Procedure: Cut fingernail
- Group B (operated):: This group will include patients who meet the same inclusion criteria as Group A. They will receive surgical treatment for claw nail by partial matrixectomy and removal of the osteophyte. They will be followed up postoperatively for 1 month, with baseline and evolutionary measurements. This group will allow to evaluate the effect of surgery on nail anatomy and symptomatology. At the end of the study, baseline and evolutionary measurements will be compared between groups to analyze the effect of surgical treatment.
  Interventions: Procedure: Exostectomy

INTERVENTIONS:
Procedure: Exostectomy — Patients diagnosed with dorsal osteophyte and experiencing pain were advised to proceed with osteophyte removal surgery during their initial visit.The surgical procedure, following protocol occurred during the second visit and involved the following steps: a 2-4 mm incision using a Beaver-64-MIS scalpel on the distal surface wall of the toe, parallel to its longitudinal axis, followed by careful osteophyte drilling; precise delineation of the osteophyte contour using a blunt elevator to prevent nailbed damage; resection executed through medial and lateral movements facilitated by a mini-Shannon drill; and finally, pressure application with a surgical spoon to extract the bone paste resulting from the drilling process.
  Groups: Group B (operated):
Procedure: Cut fingernail — Patients diagnosed with dorsal osteophyte and experiencing pain underwent nail cut fingernail
  Groups: Group A (non-operated):

SUMMARY:
This study will evaluate the usefulness of ultrasonography in detecting dorsal osteophytes associated with claw nails compared to radiographs. The hypothesis will be that the larger the size of the osteophyte, the greater the nail curvature.

Nail curvature and osteophyte height will be measured in patients with clamp nails. Nail-phalange distance will also be measured with radiography and ultrasonography.

The investigators to find a positive correlation between nail curvature and osteophyte height. Furthermore, a strong agreement is expected between both imaging techniques to measure nail-phalange distance.

Ultrasonography could constitute a safe and effective alternative to radiology for detecting dorsal osteophytes in claw nails, especially in mild cases, follow-ups or young patients.

DETAILED DESCRIPTION:
Main objective:

The investigators aim to explore the possible relationship between the degree of dorsal curvature of the nail plate and the height of the dorsal osteophyte in subungual exostosis patients before and after surgery.

Secondary objectives:

The investigators will compare the distance between the nail surface and the dorsal cortex of the distal phalanx using plain radiographs and high-resolution ultrasonography.

Materials and Methods:

This is an Interventional study patients experiencing nail pain due to clamp nails will be enrolled. Two groups will be formed depending on the presence of exostosis or not. Patients diagnosed with subungual exostosis who consent to surgery will undergo preoperative measurements. After surgery, these patients will be re-evaluated to assess the restoration of normal nail curvature values, as well as the height of the exostosis or its distance from the nail.

Measurements:

Nail curvature will be assessed using the nail curvature index, and nail height and thickness will also be measured. Dorsal osteophyte height will be assessed on radiographs and ultrasound images before and after treatment.

Expected results:

The investigators anticipate a positive correlation between dorsal osteophyte height and nail curvature. In addition, they do not expect significant differences in nail-phalange distance measurements between radiography and ultrasonography.

Conclusions:

High-resolution ultrasonography may emerge as an alternative diagnostic tool to detect subungual exostosis without exposure to ionizing radiation.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of claw nail in at least one toe.
* Pain associated with claw nail for at least 1 month.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Previous trauma or surgery on the affected toe
* Systemic diseases such as diabetes mellitus, renal insufficiency, rheumatoid arthritis
* Current or previous treatment for ingrown toenail within the last year
* Severe digital deformities (e.g. Hallux Valgus, hammer toe, claw toe)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population will be adult men and women diagnosed with painful claw nails. It is estimated to recruit 115 patients who meet the selection criteria from the podiatric consultation. The expected mean age is 45-55 years, a range consistent with the typical prevalence of this deformity. There will probably be a higher proportion of women given the greater predisposition of this sex. Participants should have nail curvatures and toenail pain of more than 1 month of evolution. Other concomitant pathologies and factors that could confound the association between osteophyte and nail curvature will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Nail-phalange distance | Pre-surgery, 2 months, 6 months.
  The measurement of the minimum distance between the dorsal cortex of the distal phalanx and the ventral aspect of the nail of the first toe will be done using lateral radiographs and longitudinal ultrasounds. Lateral radiographs capture toe images from a side angle to determine the spatial relationship between the two points, with measurements expressed in millimeters. Longitudinal ultrasounds provide real-time images to visualize this relationship, with the ultrasound transducer placed along the toe. Both methods offer vital insights into toe anatomy for medical purposes like assessing deformities, tracking injuries, or planning surgeries.

SECONDARY OUTCOMES:
Nail Curvature Index | Pre-surgery, 1 months
  The maximum height and width of the nail plate in lateral view will be measured. The curvature index will be calculated as (nail height / nail width) x 100.
Thickness of the nail plate | Pre-surgery, 1 months
  The maximum anteroposterior thickness of the nail plate in its medial part will be determined.
Dorsal Osteophyte Height | Pre-surgery, 1 months
  The height of the subungual exostosis will be measured on lateral radiographs of the distal phalanx.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guillem-Escamez, Principal Investigator — Doctorate School UCV; JAVIER FERRER TORREGROSA, Dr., Study Director — Podiatry Department, Faculty of Medicine and Health Sciences, UCV
Locations (4):
- Spain (4):
  - Enieto podologos, Logroño, La Rioja
  - Centro podológico Valencia, Valencia, València
  - Clinicas UCV, Valencia, València
  - Clinica Pasito a pasito, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vuilleumier J. [Status and problems of the physicians' assistant]. Rev Med Suisse Romande. 1979 Jul;99(7):479-81. No abstract available. French. PMID 40297
- [Result] Sano H, Shionoya K, Ogawa R. Foot loading is different in people with and without pincer nails: a case control study. J Foot Ankle Res. 2015 Aug 19;8:43. doi: 10.1186/s13047-015-0100-y. eCollection 2015. PMID 26300982
- [Result] Perez-Palma L, Manzanares-Cespedes MC, de Veciana EG. Subungual Exostosis Systematic Review and Meta-Analysis. J Am Podiatr Med Assoc. 2018 Jul;108(4):320-333. doi: 10.7547/17-102. PMID 30156888